CLINICAL TRIAL: NCT00996437
Title: An Evaluation of Intravitreal Ranibizumab for Vitreous Hemorrhage Due to Proliferative Diabetic Retinopathy
Brief Title: Intravitreal Ranibizumab for Vitreous Hemorrhage Due to Proliferative Diabetic Retinopathy (N)
Acronym: N
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEI-151; U10EY018817-03 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Vitreous Hemorrhage; Proliferative Diabetic Retinopathy
Keywords: vitreous; hemorrhage; proliferative; diabetic; retinopathy; intravitreal; ranibizumab; Lucentis; saline; vitrectomy
MeSH Terms: conditions — Vitreous Hemorrhage; Hemorrhage; Retinal Diseases | interventions — Ranibizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline Injection (Placebo Comparator): Saline injection at baseline, 4 and 8 weeks
  Interventions: Drug: Saline
- Ranibizumab (Active Comparator): Intravitreal injection of 0.5 mg ranibizumab (Lucentis™) at baseline, 4 and 8 weeks
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of 0.5 mg ranibizumab (Lucentis™) at baseline, 4 and 8 weeks
  Other Names: Lucentis
  Arms: Ranibizumab
Drug: Saline — Saline injection of 0.5mg at baseline, 4 and 8 weeks
  Arms: Saline Injection

SUMMARY:
This study is being conducted to determine if intravitreal injections of ranibizumab decrease the proportion of eyes in which vitrectomy is performed compared with saline injections in eyes presenting with vitreous hemorrhage from proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
In mild to moderate cases of vitreous hemorrhage, panretinal photocoagulation (PRP) is performed when possible to achieve regression of new vessels or at least stabilization of the neovascularization with no further growth in order to decrease the probability of subsequent vitreous hemorrhage while spontaneous absorption of the hemorrhage occurs. In cases in which the hemorrhage is too dense to apply PRP, vitrectomy is considered to remove the hemorrhage and provide a clear media for application of PRP (often as endolaser photocoagulation) as well as eliminate extensive neovascularization and relieve traction retinal detachments. Pars plana vitrectomy was introduced in the 1970s as a surgical intervention in diabetes for non-clearing vitreous hemorrhage, traction retinal detachment or very severe proliferative diabetic retinopathy (PDR). The goal of vitrectomy in such eyes is to remove the hemorrhage and provide a clear media for application of PRP (often as endolaser photocoagulation) as well as eliminate extensive neovascularization and relieve traction retinal detachments. Many advances in instrumentation and technique have resulted in a dramatic reduction in complications over the last few decades, but surgical complications remain including the following: neovascular glaucoma, retinal detachment, fibrinoid syndrome, endophthalmitis and hypotony with subsequent phthisis bulbi. Recovery for the subject can take up to 6 weeks.

Increased vascular endothelial growth factor (VEGF) levels have been demonstrated in the retina and vitreous of human eyes with diabetic retinopathy, especially PDR. VEGF has been demonstrated to increase vessel permeability by increasing the phosphorylation of tight junction proteins, and has been shown to increase retinal vascular permeability in in vivo models. Anti-VEGF therapy, therefore, may represent a useful therapeutic modality which targets the underlying pathogenesis of PDR while vitreous hemorrhage clears to facilitate the placement of PRP, potentially avoiding vitrectomy.

This study is designed to determine if intravitreal injections of ranibizumab will facilitate clearing of vitreous hemorrhage and avoidance of vitrectomy and its potential complications. Compared with a surgical intervention, use of an intravitreal agent associated with fewer vitrectomies would be preferable because of the reduced costs, reduced time to treatment, reduced intervention time, relatively low risk of side effects, and reduced recovery time. An intravitreal agent also would be a useful alternative for patients who are unwilling to undergo surgery. Furthermore, the study will determine the safety of this medication in the setting of PDR.

ELIGIBILITY:
Subject-level Criteria

Inclusion

To be eligible, the following inclusion criteria must be met:

Age >= 18 years Diagnosis of diabetes mellitus (type 1 or type 2) At least one eye meets the study eye criteria listed below Able and willing to provide informed consent.

Exclusion

A subject is not eligible if any of the following exclusion criteria are present:

A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).

A condition that, in the opinion of the investigator, would preclude subject undergoing elective vitrectomy surgery if indicated during the study.

Participation in an investigational trial that involved treatment with any drug within 30 days of randomization that has not received regulatory approval at the time of study entry.

Known allergy to any component of the study drug. Blood pressure > 180/110 (systolic above 180 or diastolic above 110). Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.

Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization.

For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 4 months.

Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 12 months of the study.

Study Eye Criteria

The subject must have at least one eye meeting all of the inclusion criteria and none of the exclusion criteria listed below.

A subject can have only one study eye. If both eyes are eligible at the time of randomization, the study eye will be selected by the investigator and subject before randomization.

The eligibility criteria for a study eye are as follows:

Inclusion

Vitreous hemorrhage causing vision impairment, presumed to be from proliferative diabetic retinopathy, and precluding completion of panretinal photocoagulation (or precluding assessment of completeness of prior PRP).

Immediate vitrectomy not required (investigator and subject are willing to wait at least 8 weeks to see if hemorrhage clears sufficiently without having to proceed to vitrectomy).

Visual acuity is light perception or better.

Exclusion

Prompt vitrectomy indicated, such as because of signs of rhegmatogenous retinal detachment or traction detachment involving the macula present on ultrasound.

Exam evidence of neovascular glaucoma, angle neovascularization, or active neovascularization of the iris (small iris tufts not an exclusion).

History of intravitreal anti-VEGF treatment for vitreous hemorrhage at any time in the past or for an indication other than vitreous hemorrhage in the past 2 months.

History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or major ocular surgery other than vitrectomy anticipated within the next 6 months following randomization.

History of vitrectomy. History of yttrium aluminum garnet capsulotomy performed within 2 months prior to randomization.

Aphakia. Uncontrolled glaucoma (in investigator's judgment). Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam R. Glassman, MS, Study Director — Jaeb Center for Health Research; Abdhish Bhavsar, MD, Study Chair — Retina Center, PA
Locations (66):
- United States (66):
  - Retinal Consultants of AZ, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retinal Consultants of Southern California Medical Group, Inc., Westlake Village, California
  - Denver Health Medical Center, Denver, Colorado
  - New England Retina Associates, PC, Trumbull, Connecticut
  - The George Washington University, Department of Ophthalmology, Washington D.C., District of Columbia
  - Retina Consultants of Southwest Florida, Fort Myers, Florida
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Magruder Eye Institute, Orlando, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Associates of Sarasota, Venice, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Georgia Retina, P.C., Atlanta, Georgia
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Retina Associates of Hawaii, Inc., Honolulu, Hawaii
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - American Eye Institute, New Albany, Indiana
  - Medical Associates Clinic, P.C., Dubuque, Iowa
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Sabates Eye Centers Research Division, Leawood, Kansas
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Retina Consultants of Delmarva, P.A., Salisbury, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - Barnes Retina Institute, St Louis, Missouri
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - Mount Sinai School of Medicine, Dept. of Ophthalmology, New York, New York
  - Retina Consultants of Western New York, Orchard Park, New York
  - Eye Care for the Adirondacks, Plattsburgh, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - University of North Carolina, Dept of Ophthalmology, Chapel Hill, North Carolina
  - Charlotte Eye Ear Nose and Throat Assoc, PA, Charlotte, North Carolina
  - Piedmont Retina Specialists, PA, Greensboro, North Carolina
  - Mid-America Retina Consultants, P.A., Kansas City, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - OSU Eye Physicians and Surgeons, LLC., Columbus, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Family Eye Group, Lancaster, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Carolina Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - West Texas Retina Consultants P.A., Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Virginia Retina Center, Leesburg, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wiconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Bhavsar AR, Torres K, Glassman AR, Jampol LM, Kinyoun JL; Diabetic Retinopathy Clinical Research Network. Evaluation of results 1 year following short-term use of ranibizumab for vitreous hemorrhage due to proliferative diabetic retinopathy. JAMA Ophthalmol. 2014 Jul;132(7):889-90. doi: 10.1001/jamaophthalmol.2014.287. No abstract available. PMID 25010170
- [Result] Diabetic Retinopathy Clinical Research Network*. Randomized clinical trial evaluating intravitreal ranibizumab or saline for vitreous hemorrhage from proliferative diabetic retinopathy. JAMA Ophthalmol. 2013 Mar;131(3):283-93. doi: 10.1001/jamaophthalmol.2013.2015. PMID 23370902
- See also: Jaeb Center for Health Research — http://www.jaeb.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab: Ranibizumab : Intravitreal injection of 0.5 mg ranibizumab (Lucentis™) at baseline, 4 and 8 weeks
- Saline Injection: Saline : Saline injection of 0.5mg at baseline, 4 and 8 weeks
Period: Overall Study
Arm/Group | Ranibizumab | Saline Injection
Started | 125 | 136
Completed | 120 | 129
Not Completed | 5 | 7
Not completed — Death | 1 | 0
Not completed — Dropped | 2 | 2
Not completed — Missed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Saline Injection | Total
Number analyzed (Participants) | 125 | 136 | 261
Age, Customized [Median (Inter-Quartile Range); unit: years] | 61 [50 to 67] | 58 [49 to 64] | 59 [50 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 70 | 135
  Male | 60 | 66 | 126
Race/Ethnicity, Customized [Number; unit: participants]
  White | 67 | 70 | 137
  African-American | 20 | 22 | 42
  Hispanic or Latino | 32 | 34 | 66
  Asian | 1 | 4 | 5
  Native Hawaiian/Other Pacific Islander | 2 | 1 | 3
  American Indian/Alaskan Native | 0 | 2 | 2
  More than one race | 2 | 1 | 3
  Unknown/not reported | 1 | 2 | 3
Diabetes Type [Number; unit: Participants]
  Type1 | 21 | 31 | 52
  Type 2 | 101 | 99 | 200
  Uncertain | 3 | 6 | 9
Duration of Diabetes (years) [Median (Inter-Quartile Range); unit: Number] | 19 [12 to 28] | 21 [16 to 27] | 20 [13 to 27]
Hemoglobin A1c [Median (Inter-Quartile Range); unit: Percentage] | 7.7 [6.7 to 8.7] | 8.0 [6.9 to 9.3] | 7.9 [6.8 to 9.0]
Pre-Existing Cardiovascular Conditions [Number; unit: Participants]
  Yes | 44 | 60 | 104
  No | 81 | 76 | 157
Pre-Existing Hypertension [Number; unit: Participants]
  Yes | 105 | 117 | 222
  No | 20 | 19 | 39
Prior panretinal photocoagulation [Number; unit: Participants]
  Yes | 62 | 78 | 140
  No | 63 | 58 | 121
Prior Treatment for Diabetic Macular Edema [Number; unit: Participants]
  Yes | 53 | 57 | 110
  No | 72 | 79 | 151
Prior treatment with anti-vascular endothelial growth factor drug for diabetic macular edema [Number; unit: Participants]
  Yes | 10 | 18 | 28
  No | 115 | 118 | 233
Lens Status (on clinical exam) [Number; unit: Participants]
  Phakic | 97 | 98 | 195
  Posterior Chamber Intraocular Lens | 28 | 38 | 66
Optical coherence tomography signal strength [Number; unit: Participants] — The Ns represent the total number of available baseline optical coherence tomography signal strengths data. Optical Coherence Tomography Signal strength is measured on a scale of 0-10 with 10 being the maximum signal strength, a greater signal strength indicates a better image.
  Participants
    =0 | 74 | 96 | 170
    > 0 | 50 | 38 | 88
    Missing/not available | 1 | 2 | 3
Ultrasound completed to assess eligibility [Number; unit: Participants]
  Yes | 62 | 62 | 124
  No | 63 | 74 | 137
Duration of vitreous hemorrhage since first documented on clinical exam [Number; unit: Participants]
  < 1month | 66 | 75 | 141
  1-3 months | 41 | 39 | 80
  4-6 months | 7 | 11 | 18
  > 6 months | 11 | 11 | 22
Median Electronic-Early Treatment Diabetic Retinopathy Visual Acuity (letter score) [Median (Inter-Quartile Range); unit: Units on a scale] — Visual Acuity was measured with the Electronic Early Treatment Study (E-ETDRS) visual acuity test. Unit of measure is based on the E-ETDRS letter score scale, 0-97, where 0 = worst and 97 = best
  Units on a scale | 34 [0 to 61] | 28 [0 to 59] | 31 [0 to 61]
Electronic Early Treatment Diabetic Retinopathy Visual Acuity Score [Number; unit: Participants] — Visual Acuity Electronic Early Treatment Study (E-ETDRS) visual acuity test (Letter Score [snellen equivalent]). Letter score and its snellen equivalent (categorical) are reported. Unit of measure is based on the E-ETDRS letter score scale, 0-97, where 0 = worst and 97 = best.
  Participants
    > 69 letter score - (20/40 or better) | 20 | 21 | 41
    68 to 49 letter score - (20/50 to 20/100) | 32 | 19 | 51
    48 to 24 letter score - (20/125 to 20/320) | 18 | 37 | 55
    23 to 1 letter score - (20/400 to 20/800-3) | 19 | 18 | 37
    Counting fingers only | 12 | 15 | 27
    Hand motion only | 19 | 20 | 39
    Light perception only | 5 | 6 | 11
    No light perception | 0 | 0 | 0
Intraocular Pressure [Median (Inter-Quartile Range); unit: mm Hg] | 15 [12 to 17] | 14 [12 to 17] | 15 [12 to 17]
Anti-platelet aggregation and anti-coagulant drugs [Number; unit: Participants] — The Ns represent concomitant medications reported throughout the study duration. Please notice that these might not be equal to the number of participants enrolled.
  Participants
    Aspirin | 50 | 57 | 107
    Other anti-platelet aggregation drugs | 19 | 21 | 40
    Anti-coagulants | 7 | 6 | 13
    NSAIDs | 15 | 15 | 30
    Not Available | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Treatment or "Failure" Defined as Vitrectomy
Description: The cumulative probabilities of vitrectomy by 16 weks (112 days) in each group were computed using the life-table method. The treatment group comparison was made using the log-rank test. Data were censored at the time point of the participant's last completed visit.
Time Frame: within 112 days of randomization
Population: The primary analysis followed the intent-to-treat principle and included all randomized eyes.
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
percentage of participants | 12 | 17
Statistical Analysis 1: Comparison: Ranibizumab vs Saline Injection; The cumulative probabilities of vitrectomy by 16 weeks in each group were computed using the life-table method. Treatment group comparisons were performed using the log-rank test. The treatment difference in cumulative probabilities and 95% confidence interval were reported; Test type: Superiority or Other; p = 0.37, Log Rank; After adjusting for potential confounding factors, time to vitrectomy remained similar between treatment groups; Treatment Difference in Cumulative Prob = 4, 95% CI 2-sided [-4 to 13]

2. Primary Outcome: Safety (Injected-related, Ocular Drug-related and Systemic Drug-related)
Time Frame: Baseline to 16 weeks
Population: Adverse events for each participants was collected throughout study duration.
Measure: Number; unit: participants
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
participants
  Endophthalmitis | 0 | 1
  Traction and/or rhegmatogeneous retinal detachment | 10 | 11
  Angle or iris neovascularization | 1 | 4
  Neovascular glaucoma | 1 | 1
  Cataract Surgery | 0 | 2
  Recurrent vitreous hemorrhage on clinical exam | 8 | 23
  Elevated Intraocular Pressure (IOP)/Glaucoma | 16 | 19
  Increase of IOP >= 10 mm Hg from baseline | 8 | 11
  IOP >= 30 mm Hg | 4 | 4
  Currently on IOP-lowering medication, not baseline | 13 | 14
  Glaucoma surgery at anytime | 0 | 0
Statistical Analysis 1: Comparison: Ranibizumab vs Saline Injection; Test type: Superiority or Other; p = 0.01, Fisher Exact — P-value corresponds with recurrent vitreous hemorrhage evaluated on clinical exam between the two treatment arms

3. Secondary Outcome: Ability to Complete Panretinal Photocoagulation (PRP) in the Absence of Vitrectomy
Description: The proportion of eyes with "complete" panretinal photocoagulation by 16 weeks in abscence of vitrectomy was computed using the life-table method and treatment groups were compared using the log-rank test.
Time Frame: within 112 days of randomization
Population: The secondary analysis followed the intent-to-treat principle and included all randomized eyes.
Measure: Number; unit: percentage of eyes
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
percentage of eyes | 44 | 31
Statistical Analysis 1: Comparison: Ranibizumab vs Saline Injection; Test type: Superiority or Other; p = 0.05, Log Rank; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [1.03 to 2.30]

4. Secondary Outcome: Extent of Vitreous Hemorrhage Measured by Optical Coherence Tomography Signal Strength
Description: Optical coherence tomography signal strength was evaluated as a potential indicator of vitreous hemorrhage density in an exploratory analysis. This analysis included only eyes with Optical Coherence Tomography (OCT) signal strength equals to 0 at baseline.
Time Frame: 4, 8 and 12 weeks
Population: This analysis followed the intent-to-treat principle
Measure: Number; unit: percentage of eyes
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
percentage of eyes
  4 week results | 40 | 28
  8 week results | 46 | 38
  12 week results | 51 | 52
Statistical Analysis 1: Comparison: Ranibizumab vs Saline Injection; Signal strength was analyzed as a composite outcome defined as OCT signal strength > = and no vitrectomy vs. OCT signal strength = 0; Test type: Superiority or Other; p = 0.87, GLM with GEE method — P-value corresponds to the 12 week visit treatment comparison; Number of subjects with baseline OCT ss=0 and OCT ss>0 and no vitrectomy at follow up. A generalized GLM with GEE was used for treatment comparisons

5. Secondary Outcome: Visual Acuity Adjusted for the Baseline Acuity Regardless of Vitrectomy Status
Description: Visual acuity was analyzed using a longitudinal mixed regression model adjusting for baseline visual acuity.Unit of measure is based on the E-ETDRS visual acuity letter score scale, 0-97, where 0 = worst and 97 = best.
Time Frame: 4, 8 and 12 weeks
Population: Number of participants with a complete 4 week visit, 8 and 12 week respectively and an available visual acuity measurement.
Measure: Mean (Standard Deviation); unit: letter scores
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
letter scores
  4 week results | 45 (30) | 42 (31)
  8 week results | 51 (30) | 47 (31)
  12 week results | 57 (27) | 49 (29)
Statistical Analysis 1: Comparison: Ranibizumab vs Saline Injection; Test type: Superiority or Other; p = .04, Mixed Models Analysis — P-value corresponds to the 12 week visit treatment comparison; Treatment comparisons were performed using a longitudinal mixed model adjusting for baseline visual acuity

6. Secondary Outcome: Visual Acuity Better Than 20/40 and no Vitrectomy Prior to the Visit
Time Frame: 4, 8 and 12 weeks
Population: This analysis followed the intent-to-treat principle. It includes all randomized eyes with a completed 4, 8 and 12 week visit respectively and an available visual acuity measure.
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
percentage of participants
  4 week results | 29 | 29
  8 week results | 36 | 33
  12 week results | 45 | 33

7. Secondary Outcome: Severe Visual Acuity Loss (Defined as <20/200)
Time Frame: 4,8 and 12 weeks
Population: Participant with a completed 4,8 and 12 week visit and an available visual acuity measurement were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
percentage of participants
  4 week results | 38 | 38
  8 week results | 30 | 35
  12 week results | 20 | 27
Statistical Analysis 1: Comparison: Ranibizumab vs Saline Injection; Test type: Superiority or Other; p = .023, Fisher Exact — P-value corresponds with the 12 week visit treatment comparison; At the each time point, treatment comparison analysis was performed using a Fisher Exact test

8. Secondary Outcome: Very Severe Visual Acuity Loss (Defined as <20/800)
Time Frame: 4,8 and 12 weeks
Population: Participants with a completed 4, 8 and 12 week visit respectively and an available visual acuity measurement were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab | Saline Injection
Number analyzed (Participants) | 125 | 136
percentage of participants
  4 week results | 20 | 25
  8 week results | 16 | 19
  12 week results | 11 | 16
Statistical Analysis 1: Comparison: Ranibizumab; Test type: Superiority or Other; p = 0.27, Fisher Exact; At each time point, treatment comparison analysis was performed using a Fisher Exact Test

ADVERSE EVENTS:
Arm/Group | Ranibizumab | Saline Injection
Serious Adverse Events (participants affected / at risk) | 13/125 | 23/136
Other Adverse Events (participants affected / at risk) | 84/125 | 94/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab (N=125) | Saline Injection (N=136)
Endophthalmitis (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 3 (3) | 4 (5)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Congestive cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic foot (Vascular disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Endocrine disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Renal Faliure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Retinal Tear (Eye disorders) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Transient ishaemic attack (Vascular disorders) | 1 (1) | 1 (1)
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab (N=125) | Saline Injection (N=136)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anterior chamber cell (Eye disorders) | 1 (1) | 0 (0)
Anterior chamber flare (Eye disorders) | 1 (1) | 0 (0)
Aphkia (Eye disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 2 (2) | 1 (1)
Ascites (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atrial fibrilliation (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Blood potasium increased (Investigations) | 1 (1) | 0 (0)
Borderline glaucoma (Eye disorders) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 5 (5) | 7 (7)
Cataract cortical (Eye disorders) | 1 (1) | 1 (1)
Cataract nuclear (Eye disorders) | 2 (3) | 0 (0)
Cataract operation complication (Eye disorders) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 2 (2) | 3 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Choroidal detachment (Eye disorders) | 0 (0) | 1 (1)
Colonic polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Conjunctival hemorrhage (Eye disorders) | 7 (11) | 7 (10)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 2 (3)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Constipation (General disorders) | 2 (2) | 1 (1)
Corneal abrasion (Eye disorders) | 2 (3) | 1 (1)
Corneal defect (Eye disorders) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Endocrine disorders) | 1 (1) | 1 (1)
Diabetic foot (Vascular disorders) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 3 (3) | 3 (3)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 3 (4) | 3 (4)
Eye pain (Eye disorders) | 14 (18) | 14 (15)
Eye pruritus (Eye disorders) | 1 (1) | 3 (6)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 9 (9)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Eye disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Endocrine disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)
Hyphaema (Eye disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Intra ocular pressure increased (Investigations) | 1 (1) | 1 (1)
Iris neovascularization (Eye disorders) | 0 (0) | 3 (3)
Irititis (Eye disorders) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 4 (4) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lung neoplasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Macular cyst (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1) | 1 (1)
Macular ischaemia (Eye disorders) | 0 (0) | 1 (2)
Mascular oedema (Eye disorders) | 1 (1) | 1 (1)
Maculopathy (Eye disorders) | 5 (5) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mammogram abnormal (Investigations) | 0 (0) | 1 (1)
Metamorphosia (Eye disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Multiple fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 8 (10) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Night blindness (Eye disorders) | 0 (0) | 1 (2)
Ocular discomfort (Eye disorders) | 2 (2) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Ocular hypertension (Eye disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 4 (5)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Parkison's disease (Nervous system disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (2) | 1 (1)
Photopsia (Eye disorders) | 4 (6) | 3 (5)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 1 (1) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal imparment (Renal and urinary disorders) | 1 (1) | 0 (0)
Retinal aneurysm (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 6 (7) | 7 (7)
Retinal disorder (Eye disorders) | 0 (0) | 2 (2)
Retinal haemorrhage (Eye disorders) | 1 (1) | 2 (2)
Retinal neovascularization (Eye disorders) | 0 (0) | 4 (5)
Retinal tear (Eye disorders) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urticaria (Immune system disorders) | 1 (1) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 8 (10) | 11 (12)
Visual acuity reduced (Eye disorders) | 6 (6) | 7 (7)
Visual field defect (Eye disorders) | 1 (2) | 0 (0)
Visual impairment (Eye disorders) | 5 (7) | 2 (2)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous disorder (Eye disorders) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 14 (15) | 11 (14)
Vitreous hemorrhage (Eye disorders) | 16 (17) | 20 (25)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No